CLINICAL TRIAL: NCT06072586
Title: A Phase 0/1 Study of BDTX-1535 in Recurrent High-Grade Glioma (HGG) and Newly Diagnosed Glioblastoma (nGBM) Participants With EGFR Alterations or Fusions Scheduled for Resection to Evaluate Central Nervous System (CNS) Penetration With PK-triggered Expansion Cohort
Brief Title: A Phase 0/1 Study of BDTX-1535 in Recurrent High-Grade Glioma (rHGG) and Newly Diagnosed Glioblastoma (nGBM) Participants With EGFR Alterations or Fusions
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Ivy Brain Tumor Center (Other); Barrow Neurological Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-20; 24-500-090-34-38 (Other: SJHMC)
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: High Grade Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: Recurrent High-Grade Glioma Participants with EGFR Alterations (Experimental): Phase 0: Cohort 1 will receive 200 mg BDTX-1535 once daily (Days 1-5). Cohort 2 will receive 400 mg BDTX-1535 three times over one week (Days 1, 3, and 5). The final dose will be administered 2-4 hours before tumor resection on Day 5.
  Phase 1: Participants will received 200 mg BDTX-1535 treatment once daily, continuously in 28-day cycles after surgery. Participants will receive BDTX-1535 until disease progression, unacceptable toxicity or death, withdrawal of consent, loss to follow-up, or study termination by the sponsor.
  Interventions: Drug: BDTX-1535
- Arm B: Recurrent High-Grade Glioma Participants with EGFR Fusion (Experimental): Phase 0: Participants will received BDTX-1535 once daily (Days 1-5). The dose level will be determined based on PK results from Arm A, unbound drug concentration in non-enhancing tumor. The final dose will be administered 2-4 hours before tumor resection on Day 5.
  Phase 1: Participants will received 200 mg BDTX-1535 treatment once daily, continuously in 28-day cycles after surgery. Participants will receive BDTX-1535 until disease progression, unacceptable toxicity or death, withdrawal of consent, loss to follow-up, or study termination by the sponsor.
  Interventions: Drug: BDTX-1535
- Arm C: Newly-Diagnosed GBM Participants with EGFR Alterations (OBD Determination) (Experimental): Phase 0: Participants in Cohort 1 will receive 200 mg of BDTX-1535 once daily for 5 days, and participants in Cohort 2 will receive 150 mg of BDTX-1535 once daily for 5 days. The final dose will be administered 2-4 hours before tumor resection on Day 5. . Participants with unmethylated MGMT promoter tumors demonstrating PK response will proceed to the Phase 1 Expansion component. The OBD will be the lowest dose that achieves the following: 9 of 12 participants show PK response and 6 of 12 participants show PD response.
  Phase 1: Participants with unmethylated MGMT promoter tumors demonstrating a PK response will continue BDTX-1535 treatment at the same dose received during Phase 0, concurrently with standard of care upfront RT, followed by adjuvant monotherapy with BDTX-1535 continuously in 28-day cycles after RT. Participants will receive BDTX-1535 until disease progression, unacceptable toxicity or death, withdrawal of consent, loss to follow-up, or study termination by the sponsor.
  Interventions: Drug: BDTX-1535 combined with radiation therapy
- Arm D: Newly-Diagnosed GBM Participants with EGFR Alterations (BDTX-1535 + RT Safety) (Experimental): Phase 0: Participants will receive the OBD of BDTX-1535 once daily for 5 days. The final dose will be administered 2-4 hours before tumor resection on Day 5. Participants with unmethylated MGMT promoter tumors demonstrating PD response will proceed to the Phase 1 Expansion component.
  Phase 1: Arm D: Participants with unmethylated MGMT promoter tumors demonstrating a PD response will continue BDTX-1535 treatment at the same dose received during Phase 0, concurrently with standard of care upfront RT, followed by adjuvant monotherapy with BDTX-1535 continuously in 28-day cycles after RT. Participants will receive BDTX-1535 until disease progression, unacceptable toxicity or death, withdrawal of consent, loss to follow-up, or study termination by the sponsor.
  Interventions: Drug: BDTX-1535 combined with radiation therapy
- Arm E: Newly-Diagnosed GBM Participants with EGFR Alterations (Stupp protocol) (Experimental): Phase 0: Participants will receive the OBD of BDTX-1535 once daily for 5 days. The final dose will be administered 2-4 hours before tumor resection on Day 5. Participants with methylated MGMT promoter tumors demonstrating PD response will proceed to the Phase 1 Expansion component.
  Phase 1: Participants with methylated MGMT promoter tumors demonstrating a PD response will continue BDTX-1535 treatment at the same dose received during Phase 0, concurrently with standard of care upfront RT and temozolomide (TMZ), followed by adjuvant BDTX-1535 combined with standard of care TMZ continuously in 28-day cycles after RT. Participants will receive BDTX-1535 until disease progression, unacceptable toxicity or death, withdrawal of consent, loss to follow-up, or study termination by the sponsor.
  Interventions: Drug: BDTX-1535 combined with temozolomide and radiation therapy

INTERVENTIONS:
Drug: BDTX-1535 — BDTX-1535 is an inhibitor of EGFR mutations
  Arms: Arm A: Recurrent High-Grade Glioma Participants with EGFR Alterations; Arm B: Recurrent High-Grade Glioma Participants with EGFR Fusion
Drug: BDTX-1535 combined with radiation therapy — During Phase 1, BDTX-1535 concurrently with standard of care upfront RT, followed by adjuvant monotherapy with BDTX-1535 continuously in 28-day cycles after RT.
  Arms: Arm C: Newly-Diagnosed GBM Participants with EGFR Alterations (OBD Determination); Arm D: Newly-Diagnosed GBM Participants with EGFR Alterations (BDTX-1535 + RT Safety)
Drug: BDTX-1535 combined with temozolomide and radiation therapy — During Phase 1, BDTX-1535 concurrently with standard of care upfront RT and TMZ, followed by adjuvant BDTX-1535 combined with standard of care TMZ continuously in 28-day cycles after RT.
  Arms: Arm E: Newly-Diagnosed GBM Participants with EGFR Alterations (Stupp protocol)

SUMMARY:
This study will administer the investigational drug, BDTX-1535 to eligible patients with recurrent high-grade glioma (HGG) and newly-diagnosed glioblastoma (nGBM). BDTX-1535 was designed to block a growth signal important to some cancers. BDTX-1535 is being tested in this study to see if it can be given safely to people who have tumors that can be dependent on that growth signal because of changes in a protein called EGFR. These gene changes are called amplifications, mutations, fusions or alterations and are found only in the tumors.

The study design includes a Phase 0 component with PK/PD-trigger for participant enrollment into an Expansion Phase 1 component. The primary objective of the Phase 0 component is to evaluate the PK endpoints of BDTX-1535. The primary objective of the Phase 1 component is to establish the safe dose of BDTX-1535 to be used in participants with a specified treatment regimen, three of which include standard of care radiotherapy for nGBM participants.

DETAILED DESCRIPTION:
The Phase 0 component will include treatment of rHGG (Arms A and B) and nGBM participants (Arms C, D, and E) with BDTX-1535 prior to a planned tumor resection. During surgery, blood, tumor, and CSF samples will be collected to measure the amount of drug that is present in the samples. Arm A includes ascending dose levels with two cohorts, and Arm C includes two dose level cohorts to determine the Optimal Biological Dose (OBD).

The Phase 1 component will include treatment in different dose regimens. Participants with tumors demonstrating PK response (Arms A, B, and C) or PD response (Arms D and E) will continue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Arms A & B: Recurrent high grade glioma (2021 WHO Grades 3 and 4), defined as participants who have progressed on or following standard therapy, which includes maximal surgical resection, temozolomide, and fractionated radiotherapy.
* Arm C, D, & E: Newly diagnosed glioblastoma (2021 WHO Grade 4), who have not received any tumor directed intervention other than biopsy or resection.
* Candidate for clinical resection of rHGG (Arms A & B) or nGBM (Arms C & D).
* Adequate archival or biopsy tissue available for testing of EGFR alterations. The tissue must have evidence of EGFR alterations including variants, fusion, and mutations with or without amplifications. rHGG participants with EGFR fusion will be solely enrolled into Arm B.
* Participants must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm.
* Provision of signed and dated, written informed consent (personally or by the legally authorized representative, if applicable) prior to any study specific procedures, sampling and analyses.
* Age ≥ 18 at time of consent
* Have a performance status (PS) of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Ability to swallow oral medications.
* Participant has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL (at time of surgery)
  * Hemoglobin ≥ 8.5 g/dL (Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.)
  * Total bilirubin ≤ 1.5 X ULN (Participants with Gilbert's syndrome with a total bilirubin ≤ 3.0 times ULN and direct bilirubin within normal limits are permitted.)
  * AST (SGOT) ≤ 3 X institutional ULN
  * ALT (SGPT) ≤ 3 X institutional ULN
  * Serum creatinine ≤ 1.5 X ULN or estimated creatinine clearance ≥ 60 mL/min (calculated using Institutional standard method)
* Participants on corticosteroids at baseline must be on stable or decreasing doses for at least 5 days prior to Day 1.
* Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
* For females of reproductive potential: use of highly effective contraception and agreement to use such a method during study participation until the end of treatment administration and for 16 weeks after the last dose of study drug.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner until the end of treatment administration and for 16 weeks after the last dose of study drug.
* Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Known allergic reactions to components of the BDTX-1535.
* Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis, as determined by the investigator.
* Known active systemic bacterial infection (requiring intravenous [IV] antibiotics or fever >38.5°C at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening of viral infection is not required for enrollment.
* Significant cardiovascular disease, including NYHA Class III or IV congestive heart failure, myocardial infarction, unstable angina, poorly controlled cardiac arrhythmias, or stroke in the preceding 6 months prior to study Day 1.
* Symptomatic or radiographic leptomeningeal disease.
* Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Concurrent use of prohibited medications: coadministration of strong CYP2C8 and CYP3A4 inhibitors and inducers with BDTX-1535. These should be discontinued 1 week or 5 half-lives (whichever is greater) prior to study Day 1. Strong inhibitors of P-gp (e.g., Amiodarone, carvedilol, dronedarone, propafenone, quinidine, ranolazine, and verapami) and BCRP (e.g., curcumin, cyclosporin A, and eltrombopag) should be used with caution. Sensitive substrates of P-gp, BCRP, and OATP should also be used with caution.
* Therapeutic intent treatment with another investigational drug or other intervention within 5 half-lives of the investigational product whichever is longer.
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v5) Grade 1 at the time of starting study treatment and patients with chronic Grade 2 unresolved toxicities may be eligible following discussion with the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Unbound BDTX-1535 Concentration in Tumor Tissue | Intraoperative
  Unbound BDTX-1535 concentration in Gd enhancing and Gd non-enhancing tumor tissue will be determined by a validated liquid chromatography-mass spectrometry (LC-MS/MS) method.
Total BDTX-1535 Concentration in Tumor Tissue | Intraoperative
  Total BDTX-1535 concentration in Gd enhancing and Gd non-enhancing tumor tissue will be determined by a validated liquid chromatography-mass spectrometry (LC-MS/MS) method.
Incidence of DLTs Observed | From day of first dose to the end of concurrent RT treatment at 10 weeks
  Considered DLTs: Hem toxicity: 8+ days ≥G4 neutropenia/febrile neutropenia; ≥G4, or ≥G3 with clinically significant bleeding, thrombocytopenia; ≥G3 anemia requiring transfusion. Non-hem lab abnormalities: Any AR ≥G3 of ALT/AST or increase in ALT/AST >3x ULN with concurrent increase in total bilirubin >2x ULN (per Hy's Law) in pt with baseline <G1 ALT/AST; Any AR ≥G3 of ALT/AST >2x baseline or 10x ULN in pt with baseline >G2 ALT/AST due to liver mets; Non-hem dose limiting toxicity ≥G3 (per Investigator; except for G3 nausea, vomiting, or diarrhea lasting <72 hrs with adequate antiemetic/supportive care; G3 fatigue or anorexia lasting <1 week; ≥G3 electrolyte abnormality lasting up to 72 hrs, isn't clinically complicated, and resolves spontaneously or responds to intervention). AR requiring dose reduction in C1, causes >2 week delay of C2, causes 8+ day dose interruption in C1.
  DLTs exclude: alopecia; lymphopenia; isolated lab changes w/o clinical sequelae or significance
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) as Assessed by NCI-CTCAE v5 | Day of first dose until 30 days after final day of participation
  AEs that occur while participants are on study treatment.
Number of Participants with Treatment-Related Adverse Events (TRAEs) as Assessed by NCI-CTCAE v5 | Day of first dose until 30 days after final day of participation
  Causality will be graded using these categories: definitely related, probably related, potentially related, unlikely to be related, and not related. Causality will be assessed by the clinician who examines and evaluates the participant based on temporal relationship and their clinical judgment. The Medical Monitor will also provide causal relationship for any Serious Adverse Events (SAEs).
Number of Participants with Abnormal Laboratory Values as Assessed per NCI-CTCAE v5 | Day of first dose until 30 days after final day of participation
  Significant changes from participant's baseline established during screening.

SECONDARY OUTCOMES:
BDTX-1535 Concentration in CSF | Intraoperative
  BDTX-1535 concentration in CSF will be determined by a validated liquid chromatography-mass spectrometry (LC-MS/MS) method.
Change in pEGFR Expression in Tumor Tissue | Baseline and intraoperative
  BDTX-1535 treated tumor tissue collected during Phase 0 surgery will be compared to archival tissue (baseline) to determine change in pEGFR expression.
Change in pERK Expression in Tumor Tissue | Baseline and intraoperative
  BDTX-1535 treated tumor tissue collected during Phase 0 surgery will be compared to archival tissue (baseline) to determine change in pERK expression.
6-Month Progression Free Survival (PFS6) Rate | From the date of Phase 0 surgery to date of disease recurrence or death, whichever occurs first, assessed up to 12 months after study completion
  PFS6 rate will be determined in participants who take at least one dose of study treatment.
Median Progression Free Survival (PFS) | From the date of Phase 0 surgery until the date of death due to any cause, assessed for up to 12 months after study completion
  Median PFS will be determined in participants with positive PK or PD response.
Median Overall Survival (OS) | From the date of Phase 0 surgery until the date of death due to any cause, assessed for up to 12 months after study completion
  Median OS will be determined in participants with positive PK or PD response.

OTHER OUTCOMES:
Total BDTX-1535 Peak Plasma Concentration (Cmax) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Bound BDTX-1535 Peak Plasma Concentration (Cmax) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Total BDTX-1535 Time to Peak Plasma Concentration (Tmax) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Bound BDTX-1535 Time to Peak Plasma Concentration (Tmax) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Total BDTX-1535 Concentration Half-Life (T1/2) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Bound BDTX-1535 Concentration Half-Life (T1/2) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Total BDTX-1535 Area Under the Plasma Concentration Versus Time Curve (AUC) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Bound BDTX-1535 Area Under the Plasma Concentration Versus Time Curve (AUC) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Total BDTX-1535 Partition Coefficient (Kp) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Unbound BDTX-1535 Partition Coefficient (Kp,uu) | Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Change in Biomarker Expression in Tumor Tissue | Baseline and intraoperative
  Tumor tissue collected during Phase 0 surgery will be compared to archival tissue (baseline) to assess fold induction change of ClCas-3, MIB-1, and pS6.
Change in Cell Signaling Pathways in Tumor Tissue | Baseline and intraoperative
  DNA, mRNA, and protein extracted from tumor tissue collected during Phase 0 surgery will be compared to those extracted from archival tissue (baseline) to examine oncogenic signaling pathways, cell cycle pathways, apoptosis pathways, and immune cell profiling using next generation sequencing analysis, single-nuclei RNA-Seq, and phospho-proteomic analysis.
Change in Single Cell State from Tumor Tissue | Baseline and intraoperative
  mRNA extracted from tumor tissue collected during Phase 0 surgery (baseline) will be compared to mRNA extracted from untreated tumor tissue collected at subsequent resections (due to recurrence) to examine changes in cell state and cellular responses.
Germline Mutation Changes in Circulating Tumor Cells (CTCs) and cell-free DNA (cfDNA) from CSF and Blood | Baseline and intraoperative
  DNA from CTCs and cfDNA extracted from CSF and blood collected during Phase 0 surgery will be compared to DNA from CTCs and cfDNA extracted from untreated CSF and blood (baseline) to examine changes in germline mutations.
Transcriptomic Changes in Circulating Tumor Cells (CTCs) from CSF and Blood | Baseline and intraoperative
  RNA from CTCs extracted from CSF and blood collected during Phase 0 surgery will be compared to RNA from CTCs extracted from untreated CSF and blood (baseline) to examine changes in the transcriptome.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Chief Scientific Officer/Director of the Ivy Brain Tumor Center
Locations (2):
- United States (2):
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ivy Brain Tumor Center Website — http://www.ivybraintumorcenter.org/